CLINICAL TRIAL: NCT01447459
Title: Effects of Educational Intervention on Long-Term Outcomes of Hospitalized Children With Asthma
Acronym: IHOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Passport Health (Industry)
Responsible Party: Principal Investigator, Tania Condurache, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Asthma IHOP - 2011
Record Dates: First submitted 2011-09-27; First posted 2011-10-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Asthma
Keywords: Asthma; Asthma Education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reinforced Education (Experimental): The caregivers of the subjects enrolled in this group will be administered two survey instruments at enrollment (t0), and again via telephone at 2 weeks (t1), 1 months (t2), and 3 months (t3) after enrollment.
  This group will also receive reinforced asthma education via telephone at 2 weeks, 1 month, and 3 months after enrollment.
  Interventions: Behavioral: Reinforced Asthma Education
- No Reinforced Education (No Intervention): The caregivers of the subjects enrolled in this group will be administered two survey instruments at enrollment (t0), and again via telephone at 2 weeks (t1), 1 month (t2), and 3 months (t3) after enrollment.
  This group will not receive reinforcing of the asthma education at 2 weeks, 1 month, and 3 months after enrollment.

INTERVENTIONS:
Behavioral: Reinforced Asthma Education — Before beginning the actual study, a board-certified Asthma Educator (AE) will prepare and administer an asthma education training session for the study personnel, including the PI, the co-investigators, and the study coordinator. The AE will also make herself available via pager for assistance with questions from the study personnel regarding asthma education.
  At the end of the administration of the phone surveys (i.e. at 2 weeks, 1 month and 3 months following enrollment), the study coordinator will provide reinforced asthma education to the caregiver via telephone for the subjects enrolled in Group A (the intervention group). The reinforced asthma education will be consistent with the asthma education training session delivered by the AE before the beginning of the study.
  Arms: Reinforced Education

SUMMARY:
The investigators hypothesize that reinforced asthma education improves long-term outcomes in children with asthma.

Specific Aims and Objectives:

1. To determine the retention rate of parental knowledge about asthma;
2. To evaluate the clinical status, quality of life and healthcare costs of children with asthma following an educational intervention.

DETAILED DESCRIPTION:
This study will be a prospective, randomized (1:1), controlled study assessing clinical status, quality of life, healthcare costs and parental retention rate of asthma knowledge for children 5 to 12 years old with asthma, following standardized asthma education versus standard education with an enhanced reinforcement of education intervention.

Group A (the intervention group) The caregivers of the subjects enrolled in this group will be administered two survey instruments at enrollment (t0), and again via telephone at 2 weeks (t1), 1 months (t2), and 3 months (t3) after enrollment. This group will also receive reinforced asthma education via telephone at 2 weeks, 1 month, and 3 months after enrollment.

Group B (the control group) The caregivers of the subjects enrolled in this group will be administered two survey instruments at enrollment (t0), and again via telephone at 2 weeks (t1), 1 month (t2), and 3 months (t3) after enrollment. This group will not receive reinforcing of the asthma education at 2 weeks, 1 month, and 3 months after enrollment.

The two survey instruments administered to the caregivers (parents/legal guardians) of the subjects enrolled in this study consist of:

1. A validated 16-item questionnaire with multiple-choice answers, assessing asthma knowledge, trigger identification and avoidance, referred to as "the Asthma Knowledge Quiz" from here on.
2. A validated 5-item questionnaire with multiple-choice answers, assessing the patient's quality of life and asthma control, referred to as "the Quality of Life/Asthma Control Test (QOL/ACT) survey" from here on.

Following enrollment and randomization, the caregiver of each subject will be administered the two survey instruments prior to discharge from the hospital.

At the end of the administration of the phone surveys (i.e. at 2 weeks, 1 month and 3 months following enrollment), the study coordinator will provide reinforced asthma education to the caregiver via telephone for the subjects enrolled in Group A (the intervention group). The reinforced asthma education will be consistent with the asthma education training session delivered by the AE before the beginning of the study.

The survey instruments will be administered to the caregiver by the study coordinator in paper form; after completion by the caregiver, the form will be saved in the subject's research binder for further data analysis. The PI or the study coordinator will determine the score for each item on the surveys, and record the scores in the subject's file, in the Asthma Knowledge Quiz Scores/Asthma Knowledge Retention Rates Form, and the Quality of Life/Asthma Control Test (QOL/ACT) Scores Form respectively.

The caregiver of each subject will be administered these two survey instruments again, via telephone, by the study coordinator, at 2 weeks, 1 month, and 3 months after enrollment. Each item and the multiple-choice answers will be literally read to the parent over the phone, and the study coordinator will record the answers to each item on the paper survey forms, which will be saved in the subject's binder for further data analysis. The PI or the study coordinator will determine the score for each survey, and record the scores in the subject's file.

A variety of statistical techniques will be used to analyze the data. The investigators will perform descriptive analyses as well as more analytic work using analysis of variance, correlation and multiple regression analysis. The investigators will use the expertise of a biostatistician to assist with accurate analysis of our data. The study will be powered to detect a significant difference in outcomes between the intervention group (group A) and the control group (group B); 25 % reduction in cost an 25% improvement in quality of life scores, following reinforced asthma education, with a 95% CI (alpha=0.05, beta=0.2, for a power of 80%). The investigators will also analyze whether there is a statistically significant correlation between the amplitude of the asthma knowledge scores (AKS) and the asthma knowledge retention rates (AKRR) on one side and the QOL/ACT scores, functional status and asthma related healthcare costs on the other side.

ELIGIBILITY:
Inclusion Criteria:

* Children age 5-12 years (eligible on or after the 5th birthday, until the day before the 13th birthday);
* Hospitalized at Norton Children's Hospital (KCH) for asthma;
* Physician diagnosis of asthma (ICD-9 codes 493.00, 493.01, 493.02, 493.10, 493.11, 493.12, 493.90, 493.91, 493.92);
* Completion of asthma education (standard of care);
* Ability of parent/legal guardian to give informed consent/research authorization, as evidenced by signing the Informed Consent Form (ICF) approved by the University of Louisville (UofL) IRB;
* Ability of subject to give informed assent for subjects equal to or older than 7 years of age, as evidenced by signing the Informed Assent Form (IAF) approved by UofL IRB.

Exclusion Criteria:

* Previous enrollment in either group of this study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Asthma Knowledge Scores (AKS) | 3 months
  The Asthma Knowledge Quiz will be administered. The higher the score (AKS), the better the knowledge of the caregiver regarding asthma, symptom recognition, trigger identification and avoidance, and medication administration. The PI or the study coordinator will calculate AKSt0, AKSt1, AKSt2, and AKSt3 (enrollment, 1 week, 2 weeks and 3 months, respectively) for each caregiver enrolled in the study. These scores will be recorded in the Asthma Knowledge Quiz Score/Asthma Knowledge Retention Rates Form for each individual subject.

SECONDARY OUTCOMES:
Asthma Knowledge Retention Rates (AKRR) | 2 weeks, 1 month, and 3 months after the initial educational intervention
  The Asthma Knowledge Retention Rates (AKRR) will be defined as the ratio between the AKS at different times during the study (i.e., t1, t2, or t3 respectively), and the AKS at baseline (AKSt0).
Quality of Life/Asthma Control Test Scores (QOL/ACT Scores) | At enrollment; 2 weeks, 1 month and 3 months after enrollment
  Quality of Life/Asthma Control (QOL/ACT) Test - each answer to 5 questions will be assigned a numeric score.
  The QOL/ACT score calculates as the sum of the scores for answers to items Q1 through Q5 for each subject. The higher the score, the better the quality of life of the patient, and the better the control achieved on asthma.
Functional Status | Enrollment; 2 weeks, 1 month and 3 months after enrollment
  Functional status will be determined by the asthma-related number of days of school absenteeism for each subject enrolled in the study. The study coordinator will collect this information from the caregivers during the follow-up phone calls at t1, t2, and t3, and record it as part of the Relevant Medical Records Form for each individual subject.
Asthma-related healthcare costs | 6 months after enrollment
  Asthma-related healthcare costs will be assessed for each subject enrolled in the study for 6 months from enrollment (t0). These costs will be calculated as the sum of the asthma-related avoidable health-care costs for the study period, including:
  * Unplanned visits to the PCP or Immediate Care Centers;
  * ED visits;
  * Hospitalizations to the pediatric ward, TCU, or PICU.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen T Condurache, M.D., Principal Investigator — University of Louisville
Locations (1):
- Norton Children's Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Background] Braman SS, Vigg A. The National Asthma Education and Prevention Program (NAEPP) guidelines: will they improve the quality of care in America? Med Health R I. 2008 Jun;91(6):166-8. No abstract available. PMID 18610803
- [Background] Bryant-Stephens T, Li Y. Community asthma education program for parents of urban asthmatic children. J Natl Med Assoc. 2004 Jul;96(7):954-60. PMID 15253327
- [Background] Bravata DM, Gienger AL, Holty JE, Sundaram V, Khazeni N, Wise PH, McDonald KM, Owens DK. Quality improvement strategies for children with asthma: a systematic review. Arch Pediatr Adolesc Med. 2009 Jun;163(6):572-81. doi: 10.1001/archpediatrics.2009.63. PMID 19487615
- [Background] Coffman JM, Cabana MD, Halpin HA, Yelin EH. Effects of asthma education on children's use of acute care services: a meta-analysis. Pediatrics. 2008 Mar;121(3):575-86. doi: 10.1542/peds.2007-0113. PMID 18310208
- [Background] Guevara JP, Wolf FM, Grum CM, Clark NM. Effects of educational interventions for self management of asthma in children and adolescents: systematic review and meta-analysis. BMJ. 2003 Jun 14;326(7402):1308-9. doi: 10.1136/bmj.326.7402.1308. PMID 12805167
- [Background] Gupta RS, Weiss KB. The 2007 National Asthma Education and Prevention Program asthma guidelines: accelerating their implementation and facilitating their impact on children with asthma. Pediatrics. 2009 Mar;123 Suppl 3:S193-8. doi: 10.1542/peds.2008-2233J. PMID 19221163
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Nicholas DB, Dell SD, Fleming-Carroll B, Selkirk EK. An evaluation of pediatric asthma educational resources. Soc Work Health Care. 2009;48(4):450-61. doi: 10.1080/00981380802589936. PMID 19396712
- [Background] McPherson AC, Glazebrook C, Forster D, James C, Smyth A. A randomized, controlled trial of an interactive educational computer package for children with asthma. Pediatrics. 2006 Apr;117(4):1046-54. doi: 10.1542/peds.2005-0666. PMID 16585298
- [Background] Murphy KR, Zeiger RS, Kosinski M, Chipps B, Mellon M, Schatz M, Lampl K, Hanlon JT, Ramachandran S. Test for respiratory and asthma control in kids (TRACK): a caregiver-completed questionnaire for preschool-aged children. J Allergy Clin Immunol. 2009 Apr;123(4):833-9.e9. doi: 10.1016/j.jaci.2009.01.058. PMID 19348922
- [Background] Lara M, Rosenbaum S, Rachelefsky G, Nicholas W, Morton SC, Emont S, Branch M, Genovese B, Vaiana ME, Smith V, Wheeler L, Platts-Mills T, Clark N, Lurie N, Weiss KB. Improving childhood asthma outcomes in the United States: a blueprint for policy action. Pediatrics. 2002 May;109(5):919-30. doi: 10.1542/peds.109.5.919. PMID 11986457
- [Background] Taggart VS, Zuckerman AE, Sly RM, Steinmueller C, Newman G, O'Brien RW, Schneider S, Bellanti JA. You Can Control Asthma: evaluation of an asthma education program for hospitalized inner-city children. Patient Educ Couns. 1991 Feb;17(1):35-47. doi: 10.1016/0738-3991(91)90049-b. PMID 1997997
- [Background] Wang LY, Zhong Y, Wheeler L. Direct and indirect costs of asthma in school-age children. Prev Chronic Dis. 2005 Jan;2(1):A11. Epub 2004 Dec 15. PMID 15670464
- [Background] Asthma prevalence, Health Care Use and Mortality, 2002. National Center for Health Statistics, Health Data for All Ages (HDAA). http://www.cdc.gov/nchs/products/pubs/pubd/hestats/asthma/asthma.htm.
- See also: Kosair Charities Pediatric Clinical Research Unit — https://louisville.edu/medschool/pediatrics/research/kcpcru